CLINICAL TRIAL: NCT00340899
Title: Biological Markers of Disease in the Prediction of Preterm Delivery, Preeclampsia and Intra-Uterine Growth Restriction: A Longitudinal Study
Brief Title: Biological Markers of Disease in the Prediction of Preterm Delivery, Preeclampsia and Intra-Uterine Growth Retardation: A Longtitudinal Study
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997067; OH97-CH-N067
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Prenatal Care; Premature Birth
Keywords: Perinatal Mortality; Perinatal Morbidity; Preterm Birth; Pregnancy Complications; Pregnancy; Natural History
MeSH Terms: conditions — Premature Birth; Perinatal Death; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women with gestational age between 6 and 22 weeks

SUMMARY:
Preterm delivery, preeclampsia and intrauterine growth restriction are leading causes of perinatal morbidity and mortality. Efforts to treat these syndromes have not been effective, most likely becuase these obstetric complications are the clinical expression of adaptive mechanisms of host defense developed in response to pathologic insults. Since the ultimate pathologic basis of disease is unclear, therapy for these syndromes has been largely directed at symptoms, which appear late in the development of the disease. The main purpose of this study is to perform an early and comprehensive exploration of maternal and fetal factors that predict the subsequent develpment of these obstetrice complications, so that early medical interventions may be tested in patients at high and low risk for adverse perinatal outcome.

DETAILED DESCRIPTION:
Preterm delivery, preeclampsia and intrauterine growth restriction are leading causes of perinatal morbidity and mortality. Efforts to treat these syndromes have not been effective, most likely because these obstetric complications are the clinical expression of adaptive mechanisms of host defense developed in response to pathologic insults. Since the ultimate pathologic basis of disease is unclear, therapy for these syndromes has been largely directed at symptoms, which appear late in the development of the disease. The main purpose of this study is to perform an early and comprehensive exploration of maternal and fetal factors that predict the subsequent development of these obstetric complications, so that early medical interventions may be tested in patients at high and low risk for adverse perinatal outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Gestational age between 6 and 22 weeks for the first visit based on the patient s last menstrual period as reported by the patient.
* High risk group: presence of specific risk factors for preterm delivery, pregnancy-induced hypertension or intrauterine growth retardation.
* Low risk group: normal pregnancy with no risk factors for preterm delivery, pregnancy-induced hypertension or intrauterine growth retardation (control population, selected between 6 and 22 weeks at the prenatal care clinic). The rationale to include this group is that 50-70% of preterm deliveries occur in patients without risk factors for preterm birth.
* Consent to participate in the study.
* Patient should be able to attend each Perinatal Research Center for prenatal care and participation in this study.

EXCLUSION CRITERIA:

* Preterm labor, preterm PROM, preeclampsia or impaired fetal growth at the time of recruitment.
* Any maternal or fetal condition that requires termination of pregnancy.
* Known major fetal anomaly or fetal demise.
* Active vaginal bleeding.
* Multifetal pregnancy with greater than or equal to 3 fetuses.
* Serious medical illness (renal insufficiency, congestive heart disease, chronic respiratory insufficiency, etc).
* Severe chronic hypertension (requiring medication).
* Asthma requiring systemic steroids.
* Patient requiring anti-platelet or non-steroidal anti-inflammatory drugs.
* Active hepatitis.
* Lack of consent.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant women attending prenatal clinics
Sampling Method: Non-Probability Sample
Enrollment: 19134 (Actual)
Dates: Start 1997-12-04 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Preterm delivery | Ongoing
  Preterm delivery will be classified according to the immediate clinical antecedent of delivery (spontaneous preterm labor with intactmembranes, preterm premature rupture of membranes and pretermdelivery for maternal or fetal indications).
Preeclampsia | Ongoing
  Preeclampsia will be defined according to the following criteria:-Systolic blood pressure greater than or equal to 140 mmHg and/or diastolic blood pressure greater than or equal to 90 mmHg on twooccasions greater than or equal to 6 hours apart.-Proteinuria greater than or equal to 300 mg/24 hr or freater than or equal to 2+ (dipstick) on two occasions greater than or equal to 6 hours apart.-The diagnosis of severe preeclampsia will be made in the presence of any of the following: blood pressure greater than or equal to 160 mmHg (systolic) or greater than or equal to 110 (diastolic) on at least two occasions, proteinuria greater than or equal to 5 gr /24 hr, pulmonary edema, thrombocytopenia, oliguria, neurologic symptoms(headache, visual disturbances, persistent hyperreflexia, upperabdominal pain and HELLP syndrome). Eclampsia will be diagnosed if convulsions develop.
Intrauterine growth restriction | Ongoing
  Intrauterine growth retardation / small for gestational age infantA small for gestational age fetus will be considered that with a birth weight which is below the 10th percentile for gestational age. Additional cutoffs (5th and 3rd percentile) will also be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Sotero del Rio Hospital, Santiago, Chile

REFERENCES:
- [Background] Pollack RN, Divon MY. Intrauterine growth retardation: definition, classification, and etiology. Clin Obstet Gynecol. 1992 Mar;35(1):99-107. doi: 10.1097/00003081-199203000-00015. No abstract available. PMID 1544253
- [Background] Romero R, Mazor M, Wu YK, Sirtori M, Oyarzun E, Mitchell MD, Hobbins JC. Infection in the pathogenesis of preterm labor. Semin Perinatol. 1988 Oct;12(4):262-79. No abstract available. PMID 3065940
- [Background] Harding JE, Owens JA, Robinson JS. Should we try to supplement the growth retarded fetus? A cautionary tale. Br J Obstet Gynaecol. 1992 Sep;99(9):707-9. doi: 10.1111/j.1471-0528.1992.tb13866.x. No abstract available. PMID 1343567